CLINICAL TRIAL: NCT04817644
Title: A Trial Investigating Semaglutide and SNAC Concentrations in Breastmilk Following Administration of Multiple Doses of Oral Semaglutide in Healthy, Lactating Females
Brief Title: A Research Study to See How Much Semaglutide and SNAC is in the Milk of Healthy, Breastfeeding Women Taking Semaglutide Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4669; U1111-1253-4467 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral semaglutide (Experimental): All participants will receive oral semaglutide once daily for a total of 10 days: 3 mg for 5 days followed by 7 mg for 5 days.
  Interventions: Drug: Oral semaglutide

INTERVENTIONS:
Drug: Oral semaglutide — Oral semaglutide once daily for a total of 10 days

SUMMARY:
Participants in the study, will receive the study drug once daily for 10 days in tablet form for oral (by mouth) intake. On day 1 to 5 the tablet will contain 3 mg semaglutide, and on day 6-10 the tablet will contain 7 mg semaglutide.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, female subjects who have given birth at least 3 months prior to screening and who breastfeed (breastfeeding is defined by feeding the baby milk produced by the mother. Using a breast pump to collect milk and subsequently feeding it to the baby by bottle, is also defined as breastfeeding ) their infant to an extent, where the majority of the infant's total energy intake is from breastfeeding and sufficient milk is produced to fulfil the trial requirements, as judged by the investigator.
* Agree to abstain from breastfeeding their infant from first dose of oral semaglutide to the "End of trial" visit (total of 47 days) to avoid potentially exposing their child to semaglutide and SNAC.
* The breastfed infant is able to feed from a bottle (expenses related to alternative infant nutrition during trial participation will be covered by Novo Nordisk) prior to screening.
* Age above or equal to 18 years at the time of agreement to take part.
* Body mass index (BMI) between 20.0 and 32.4 kg/m^2 (both inclusive).

Exclusion Criteria:

* Female who is pregnant or intends to become pregnant or is of child-bearing potential and not using an effective contraceptive method.
* Glycated haemoglobin (HbA1c) greater than or equal to 6.5 % (48 mmol/mol) at screening.
* Presence of clinically significant gastrointestinal disorders or symptoms of gastrointestinal disorders potentially affecting absorption of drugs or nutrients, as judged by the investigator.
* History (as declared by the subject or reported in the medical records) of major surgical procedures involving the stomach potentially affecting absorption of trial products (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery).
* Personal or first degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma (as declared by the subject or reported in the medical records).
* Presence or history (as declared by the subject or reported in the medical records) of malignant neoplasm within 5 years prior to the day of screening (basal or squamous cell skin cancer, or any carcinoma in-situ is allowed).
* Presence or history (as declared by the subject or reported in the medical records) of pancreatitis (acute or chronic).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Area under the semaglutide milk concentration-time curve during a dosing interval after the 10th dosing (AUC0-24h,sema,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  nmol*h/L
Area under the salcaprozate sodium (SNAC) milk concentration-time curve during a dosing interval after the 10th dosing (AUC0-24h,SNAC,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng*h/mL

SECONDARY OUTCOMES:
Average semaglutide milk concentration during a dosing interval after the 10th dosing (Cavg,sema,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  nmol/L
Maximum semaglutide milk concentration during a dosing interval after the 10th dosing (Cmax,sema,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  nmol/L
Minimum semaglutide milk concentration during a dosing interval after the 10th dosing (Cmin,sema,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  nmol/L
Time to maximum semaglutide milk concentration during a dosing interval after the 10th dosing (tmax,sema,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  Hours
Estimated daily infant semaglutide dose | From 0 to 24 hours after the 10th dosing (day 10)
  mg/kg/day
Relative daily infant semaglutide dose | From 0 to 24 hours after the 10th dosing (day 10)
Average SNAC milk concentration during a dosing interval after the 10th dosing (Cavg,SNAC,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Maximum SNAC milk concentration during a dosing interval after the 10th dosing (Cmax,SNAC,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Minimum SNAC milk concentration during a dosing interval after the 10th dosing (Cmin,SNAC,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Time to maximum SNAC milk concentration during a dosing interval after the 10th dosing (tmax,SNAC,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  hours
Estimated daily infant SNAC dose | From 0 to 24 hours after the 10th dosing (day 10)
  ng/kg/day
Relative daily infant SNAC dose | From 0 to 24 hours after the 10th dosing (day 10)
Area under the SNAC metabolite E494 milk concentration-time curve during a dosing interval after the 10th dosing (AUC0-24h,E494,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng*h/mL
Average SNAC metabolite E494 milk concentration during a dosing interval after the 10th dosing (Cavg,E494,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Maximum SNAC metabolite E494 milk concentration during a dosing interval after the 10th dosing (Cmax,E494,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Minimum SNAC metabolite E494 milk concentration during a dosing interval after the 10th dosing (Cmin,E494,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Time to maximum SNAC metabolite E494 milk concentration after the 10th dosing (tmax,E494,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  hours
Estimated daily infant SNAC metabolite E494 dose | From 0 to 24 hours after the 10th dosing (day 10)
  ng/kg/day
Area under the SNAC metabolite E506 milk concentration-time curve during a dosing interval after the 10th dosing (AUC0-24h,E506,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng*h/mL
Average SNAC metabolite E506 milk concentration during a dosing interval after the 10th dosing (Cavg,E506,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Maximum SNAC metabolite E506 milk concentration during a dosing interval after the 10th dosing (Cmax,E506,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Minimum SNAC metabolite E506 milk concentration during a dosing interval after the 10th dosing (Cmin,E506,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Time to maximum SNAC metabolite E506 milk concentration after the 10th dosing (tmax,E506,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  hours
Estimated daily infant SNAC metabolite E506 dose | From 0 to 24 hours after the 10th dosing (day 10)
  ng/kg/day
Area under the SNAC metabolite E1245 milk concentration-time curve during a dosing interval after the 10th dosing (AUC0-24h,E1245,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng*h/mL
Average SNAC metabolite E1245 milk concentration during a dosing interval after the 10th dosing (Cavg,E1245,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Maximum SNAC metabolite E1245 milk concentration during a dosing interval after the 10th dosing (Cmax,E1245,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Minimum SNAC metabolite E1245 milk concentration during a dosing interval after the 10th dosing (Cmin,E1245,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Time to maximum SNAC metabolite E1245 milk concentration after the 10th dosing (tmax,E1245,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  hours
Estimated daily infant SNAC metabolite E1245 dose | From 0 to 24 hours after the 10th dosing (day 10)
  ng/kg/day
Area under the SNAC metabolite E1246 milk concentration-time curve during a dosing interval after the 10th dosing (AUC0-24h,E1246,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng*h/mL
Average SNAC metabolite E1246 milk concentration during a dosing interval after the 10th dosing (Cavg,E1246,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Maximum SNAC metabolite E1246 milk concentration during a dosing interval after the 10th dosing (Cmax,E1246,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Minimum SNAC metabolite E1246 milk concentration during a dosing interval after the 10th dosing (Cmin,E1246,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Time to maximum SNAC metabolite E1246 milk concentration in milk after the 10th dosing (tmax,E1246,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  hours
Estimated daily infant SNAC metabolite E1246 dose | From 0 to 24 hours after the 10th dosing (day 10)
  ng/kg/day
Area under the SNAC metabolite E1247 milk concentration-time curve during a dosing interval after the 10th dosing (AUC0-24h,E1247,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng*h/mL
Average SNAC metabolite E1247 milk concentration during a dosing interval after the 10th dosing (Cavg,E1247,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Maximum SNAC metabolite E1247 milk concentration during a dosing interval after the 10th dosing (Cmax,E1247,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Minimum SNAC metabolite E1247 milk concentration during a dosing interval after the 10th dosing (Cmin,E1247,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Time to maximum SNAC metabolite E1247 milk concentration after the 10th dosing (tmax,E1247,D10,milk) | From 0 to 24 hours after the 10th dosing (day 10)
  hours
Estimated daily infant SNAC metabolite E1247 dose | From 0 to 24 hours after the 10th dosing (day 10)
  ng/kg/day
Area under the semaglutide plasma concentration-time curve during a dosing interval after the 10th dosing (AUC0-24h,sema,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  nmol*h/L
Maximum semaglutide plasma concentration during a dosing interval after the 10th dosing (Cmax,sema,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  nmol/L
Time to maximum semaglutide plasma concentration during a dosing interval after the 10th dosing (tmax,sema,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  hours
Area under the SNAC plasma concentration-time curve during a dosing interval after the 10th dosing (AUC0-24h,SNAC,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  ng*h/mL
Maximum SNAC plasma concentration during a dosing interval after the 10th dosing (Cmax,SNAC,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Time to maximum SNAC plasma concentration during a dosing interval after the 10th dosing (tmax,SNAC,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  hours
Area under the SNAC metabolite E494 plasma concentration-time curve during a dosing interval after the 10th dosing (AUC0-24h,E494,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  ng*h/mL
Maximum SNAC metabolite E494 plasma concentration during a dosing interval after the 10th dosing (Cmax,E494,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Time to maximum SNAC metabolite E494 plasma concentration during a dosing interval after the 10th dosing (tmax,E494,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  hours
Area under the SNAC metabolite E506 plasma concentration-time curve during a dosing interval after the 10th dosing (AUC0-24h,E506,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  ng*h/mL
Maximum SNAC metabolite E506 plasma concentration during a dosing interval after the 10th dosing (Cmax,E506,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Time to maximum SNAC metabolite E506 plasma concentration during a dosing interval after the 10th dosing (tmax,E506,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  hours
Area under the SNAC metabolite E1245 plasma concentration-time curve during a dosing interval after the 10th dosing (AUC0-24h,E1245,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  ng*h/mL
Maximum SNAC metabolite E1245 plasma concentration during a dosing interval after the 10th dosing (Cmax,E1245,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Time to maximum SNAC metabolite E1245 plasma concentration during a dosing interval after the 10th dosing (tmax,E1245,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  hours
Area under the SNAC metabolite E1246 plasma concentration-time curve during a dosing interval after the 10th dosing (AUC0-24h,E1246,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  ng*h/mL
Maximum SNAC metabolite E1246 plasma concentration during a dosing interval after the 10th dosing (Cmax,E1246,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Time to maximum SNAC metabolite E1246 plasma concentration during a dosing interval after the 10th dosing (tmax,E1246,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  hours
Area under the SNAC metabolite E1247 plasma concentration-time curve during a dosing interval after the 10th dosing (AUC0-24h,E1247,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  ng*h/mL
Maximum SNAC metabolite E1247 plasma concentration during a dosing interval after the 10th dosing (Cmax,E1247,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  ng/mL
Time to maximum SNAC metabolite E1247 plasma concentration during a dosing interval after the 10th dosing (tmax,E1247,D10,plasma) | From 0 to 24 hours after the 10th dosing (day 10)
  hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - ICON Early Phase Services, LLC, San Antonio, Texas
  - ICON-Salt Lake City, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com